CLINICAL TRIAL: NCT03584659
Title: Patient-reported Outcomes in Bladder Cancer; a Multicentre Randomized Controlled Trial: The iBLAD Study
Brief Title: Patient-reported Outcomes in Bladder Cancer
Acronym: iBLAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Herlev Hospital (Other); Danish Cancer Society (Other); Aalborg University Hospital (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Helle Pappot, Clinical Oncologist, Consultant, DMSc, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: iBLAD2018
Record Dates: First submitted 2018-06-21; First posted 2018-07-12 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Bladder Cancer; Urothelial Carcinoma
Keywords: Patient-reported outcomes; Electronic reporting of symptoms; Immunotherapy; Chemotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): This arm will continue standard procedure regarding side effect registration and handling
- PRO (Experimental): This arm will be assigned to intervention by weekly electronic reporting of side effects and quality of life. A specifically developed alert-algorithm will in real-time guide both patient and alert clinical staff if symptoms are increasing or quality of life is deteriorating.
  Interventions: Device: Electronic patient-reported outcomes

INTERVENTIONS:
Device: Electronic patient-reported outcomes — Weekly reporting of patient-reported outcomes for closer contact between patient and clinic between treatment cycles.
  Other Names: Alert-algorithm; Real-time guidance of patients when symptom reporting; Alerts to clinical staff
  Arms: PRO

SUMMARY:
Electronic reporting of patient-reported outcomes with alert algorithm will be tested in a randomized trial in bladder cancer patients undergoing chemo- or immunotherapy. The clinical endpoints will be:

* Quality of life
* Completion of treatment
* Hospital admission
* Dose reductions
* Survival

DETAILED DESCRIPTION:
Bladder cancer is in Europe the 4th most incident cancer among men and the 7th most frequent cause of cancer death. Many patients will receive chemo- or immunotherapy in either the neoadjuvant setting or for recurrent or metastatic disease. The registration and handling of side effect is crucial in bladder cancer treatment, since the missing identification and insufficient treatment of such can lead to incomplete treatment and thereby decreased effect. It is therefore of utmost importance to develop new tools which can increase identification of the side effects and improve treatment to secure the best life expectancies for these patients.

This study will in a randomized trial using PRO-CTCAE™ questions, EORTC QLQ-C30 + QLQ-BLM30 in one arm versus standard procedure regarding side effect registration and handling in the other arm, test the effect of electronic reporting of side-effects and quality of life with a specifically developed alert-algorithm. Both study arms will include chemotherapy and immunotherapy patients as standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Urothelial carcinoma
* Initiating chemo- or immunotherapy
* No serious cognitive deficits
* Read and understand Danish
* Assigned electronic communication with health services with "E-boks"

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Rate of completion of treatment | Within the first 6 months of treatment
  Registration of whether patients complete the planned treatment and if not if the cessation was preventable.
Hospital admission | Within the first 6 months of treatment
  Registration of whether patients by closer contact to clinic between visits can decrease the rate of hospital admissions for preventable causes during treatment.

SECONDARY OUTCOMES:
Quality of life questionnaires EORTC QLQ-C30 (general quality of life questionnaire) and EORTC QLQ-BLM30(quality of life questionnaire specifically for muscle-invasive bladder cancer patients) | Within the first 6 months of treatment
  Registration of differences in quality of life between the two arms in the study. EORTC QLQ-C30(scale range 0-100, a higher score indicating better quality of life) and QLQ-BLM30(scale range 0-100, a higher score indicating increase in symptom burden) will be used for as quality of life measurement. The scores will be presented graphically in separate figures. The EORTC QLQ-BLM30 cannot be applied without the QLQ-C30, hence the aggregation of measures in the present outcome measure category.
  Differences between the two arms will be tested using t-test and analysis of covariance (ANCOVA).
Overall survival measured from time of study initiation to death | Analysis will be made up to 2 years after study completion
  Differences in median overall survival and analysis of survival differences between the intervention-arm and the standard of care arm. The analysis will be carried out with log-rank analysis and Kaplan-Meier curves. The analysis will be carried out separately for chemotherapy and immunotherapy recipients.
Dose-reductions | Within the first 6 months of treatment
  Registration of differences in number of dose reductions of chemotherapy between the two arm in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Gry Assam Taarnhøj, MD, Principal Investigator — Department of Oncology, Copenhagen University Hospital, Rigshospitalet, Denmark
Locations (4):
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Department of Oncology, Rigshospitalet, Copenhagen
  - Department of Oncology, Herlev
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taarnhoj GA, Johansen C, Carus A, Dahlrot RH, Dohn LH, Hjollund NH, Knudsen MB, Tolver A, Lindberg H, Pappot H. The iBLAD study: patient-reported outcomes in bladder cancer during oncological treatment: a multicenter national randomized controlled trial. J Patient Rep Outcomes. 2023 Oct 9;7(1):99. doi: 10.1186/s41687-023-00640-5. PMID 37812306